CLINICAL TRIAL: NCT04240210
Title: SymITA: Switch to DRV/COB/FTC/TAF From Integrase Containing Regimens to Evaluate Changes in Tolerability/Adherence
Brief Title: Integrase Regimen Switch to Symtuza to Increase Tolerability/Adherence (SYMita)
Acronym: SymITA
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of eligible enrollees/ Halted by Primary Sponsor
Sponsor: Midland Research Group, Inc. (Other)
Collaborators: Janssen Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TMC114FD2HTX4005
Record Dates: First submitted 2020-01-06; First posted 2020-01-27 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Human Immunodeficiency Virus
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — symtuza

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- To assess degree of adherence to ART in a real world seeting. (No Intervention): Part I of the study is a Cohort Survey of HIV+ outpatient clinic patients currently receiving ART to assess medication adherence and tolerability by determining a change in adherence and tolerability from baseline to 4 months, measured by standardized patient reported outcome and adherence surveys
- Potential changes in ART adherence when switced to Symtuza. (Experimental): Part 2 of the study is a prospective cohort analysis of change in adherence, tolerability and safety of subjects who reports poor adherence to ART due to intolerance/side effects from integrase inhibitor containing regimens when they are switched to DRV/COB/FTC/TAF and monitored for 4 months.
  Interventions: Drug: Symtuza

INTERVENTIONS:
Drug: Symtuza — The study is a prospective cohort analysis of change in adherence, tolerability and safety of subjects who reports poor adherence to ART due to intolerance/side effects from integrase inhibitor containing regimens when they are switched to DRV/COB/FTC/TAF and monitored for 4 months.
  Arms: Potential changes in ART adherence when switced to Symtuza.

SUMMARY:
Darunavir/cobicistat/emtricitabine/tenofovir alafenamide (DRV/COB/FTC/TAF) is a coformulated STR, is the only protease inhibitor based STR, and is noted for its high tolerability3. These traits have the potential to improve adherence in patients who have intolerance to the integrase inhibitor class. We propose a two part study design to evaluate if patients who have suboptimal adherence due to integrase inhibitor intolerance may better tolerate Symtuza and subsequently have improved adherence.

DETAILED DESCRIPTION:
With the advent of anti-retroviral therapy, HIV transformed into a manageable chronic disease for patients who were able to obtain medications, provided they could remain adherent to them. When single tablet regimens (STR) became available, adherence to HIV medications was made easier for many patients. However even years after STR became available, 38% of patients reported they do not maintain optimal adherence to their HIV medications. While there are many factors that contribute to this problem, medication intolerance contributes to suboptimal adherence for many patients

Darunavir/cobicistat/emtricitabine/tenofovir alafenamide (Symtuza) is a coformulated STR, is the only protease inhibitor based STR, and is noted for its high tolerability. This trait has the potential to improve adherence in patients who have intolerance to the integrase inhibitor class. We are not aware of any studies that have examined this potential and find that information gap worth investigating.

We propose a two part study design to evaluate if patients who have suboptimal adherence due to integrase inhibitor intolerance may have better tolerability to Symtuza and subsequently have improved adherence.

The initial portion of the study will consist of a self-administered adherence survey offered over a 4 month period to established patients at Midland Medical Center who are HIV+, regardless of disease state or regimen. Subjects who self-identify as non-adherent due to tolerability issues will be screened for enrollment in the primary study. Subjects found to be non-adherent due to other issues will be referred back to their provider.

Subjects who are referred for screening who are on an integrase inhibitor and who do not have a contraindication will be enrolled, will complete a Patient Reported Outcome survey (PRO) to assess side effects/quality of life, and switched to Symtuza. Subjects who are not enrolled in the study will be referred back to their provider to address the issues with tolerance and adherence.

Subjects will be followed for 4 months. During that period, they will be brought back for evaluation at the end of the first month and the end of the fourth month. At those evaluations, they will again complete the PRO and adherence surveys to assess tolerability and adherence. At the evaluations, they will also be monitored for safety and effectiveness via physical exams and laboratory studies (Complete Blood Count, Complete Metabolic Panel, Urinalysis, CD4 panel, HIV1 Quantitative viral load).

The de-identified laboratory and survey results from the baseline and subsequent assessments will be turned over to a statistician to evaluate changes in adherence, tolerability, effectiveness, and safety.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age.
* HIV positive receiving ART of any type.
* Currently on an integrase containing regimen AND Reports non-adherent due to medication intolerance.
* GFR≥30mL/min.
* AST/ALT ≤ 3 times upper limit of normal. (AST- U/L 10-40), (ALT- U/L 9-46)
* Total bilirubin of ≤1.5 mg/dL.

Exclusion Criteria:

* Known resistance to darunavir or tenofovir
* Known intolerance to Symtuza or its components
* Current pregnancy
* Requires continued use of any of the agents in table 6.2.3.2.4
* Cirrhosis, regardless of compensation status
* Active, serious infections within 30 days of baseline
* History of malignancy within 5 years of baseline, except cutaneous Kaposi's sarcoma, basal cell or resected non-invasive cutaneous squamous cell carcinoma
* Life expectancy of less than a year
* Participation in any other investigation study 30 days prior to enrollment

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-09-17 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Part 1 of the study is a cohort survey of change in adherence, tolerability and safety of subjects who report poor adherence to ART due to intolerance/side effects from integrase inhibitor containing regimens. | 4 months
  To evaluate trends and patterns in subjects who report sub-optimal adherence, analyzed by intention to treat with Integrase Inhibitor based Antiretroviral containing regimens, based upon the subjects completion of the Midland ART Adherence Survey (MAAS)

SECONDARY OUTCOMES:
To determine potential changes in ART adherence in subjects who report sub-optimal adherence due to side effects from integrase containing regimens after switching to Symtuza. | 4 months
  Sub-optimal adherence will be determined by comparing the study subjects completed Midland ART Adherence Survey at the week 4 visit to the week 16 visit to the number of the investigational product (Symtuza) tablets that are counted at week 4 visit and week 16 visit.
  Each dispensed bottle of IP (Symtuza) will contain 30 tablets.
To evaluate the tolerability of switching from an integrase inhibitor containing regimen to Symtuza. | 4 months
  We will be using the standardized Patient Reported Outcomes (PRO) questionnaire to determine a percentage of subjects who report suboptimal adherence due to tolerance issues/side effects and those who report suboptimal adherence due to reasons other than tolerance issues/side effects.
Safety and efficacy of switching from integrase inhibitor containing regimen to Symtuza as determined by the proportion of subjects with virologic failure, a change in laboratory parameters and change in CD4 cell count from baseline. | 4 months
  1. We will be looking at the proportion of subjects that have an HIV-1 RNA ≥ 50 copies/mL at baseline and at week 16 and comparing them to the subjects level of ART adherence.
  2. There will be an assessment of whether or not there are any significant laboratory changes in subjects serum Creatinine- (0.70-1.33 mg/dL) , AST- (10-35 u/L) and ALT-(9-46 u/L) when compared to week 16 from the baseline evaluation.
  3. We will compare any laboratory changes in the subjects Absolute CD4+ cell count- (490-1740 cells/uL) along with the % of CD4 cells- (30-61%) from the subjects week 16 laboratory levels to the baseline assessment by using the study site determined laboratory.
To evaluate for potential weight loss when switching from integrase inhibitor containing regimen to Symtuza. | 4 months
  There will be an assessment of the subjects weight in kilograms- (kg) from the initial baseline visit to the week 16 visit with recorded BMI.
  Initial subjects Body Mass Index (BMI) will be assessed by using the formula: weight (kg) / [height (m)]2
  The World Health Organization's (WHO) recommended body weight based on BMI values for adults will be referenced.
  Category BMI range - kg/m2 Severe Thinness < 16 Moderate Thinness 16 - 17 Mild Thinness 17 - 18.5 Normal 18.5 - 25 Overweight 25 - 30 Obese Class I 30 - 35 Obese Class II 35 - 40 Obese Class III > 40

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Ciesielski, MD, Principal Investigator — Midland Research Group
Locations (1):
- Midland Research Group, Inc, Oakland Park, Florida, United States

REFERENCES:
- [Background] Ortego C, Huedo-Medina TB, Llorca J, Sevilla L, Santos P, Rodriguez E, Warren MR, Vejo J. Adherence to highly active antiretroviral therapy (HAART): a meta-analysis. AIDS Behav. 2011 Oct;15(7):1381-96. doi: 10.1007/s10461-011-9942-x. PMID 21468660
- [Background] Robbins RN, Spector AY, Mellins CA, Remien RH. Optimizing ART adherence: update for HIV treatment and prevention. Curr HIV/AIDS Rep. 2014 Dec;11(4):423-33. doi: 10.1007/s11904-014-0229-5. PMID 25304006
- [Background] Orkin C, Molina JM, Negredo E, Arribas JR, Gathe J, Eron JJ, Van Landuyt E, Lathouwers E, Hufkens V, Petrovic R, Vanveggel S, Opsomer M; EMERALD study group. Efficacy and safety of switching from boosted protease inhibitors plus emtricitabine and tenofovir disoproxil fumarate regimens to single-tablet darunavir, cobicistat, emtricitabine, and tenofovir alafenamide at 48 weeks in adults with virologically suppressed HIV-1 (EMERALD): a phase 3, randomised, non-inferiority trial. Lancet HIV. 2018 Jan;5(1):e23-e34. doi: 10.1016/S2352-3018(17)30179-0. Epub 2017 Oct 6. PMID 28993180

DOCUMENTS (2):
  • Study Protocol (2019-12-17): https://cdn.clinicaltrials.gov/large-docs/10/NCT04240210/Prot_001.pdf
  • Informed Consent Form (2019-12-17): https://cdn.clinicaltrials.gov/large-docs/10/NCT04240210/ICF_000.pdf